CLINICAL TRIAL: NCT04143126
Title: Cognitive Enhancement for Persistent Negative Symptoms in Schizophrenia
Brief Title: Promoting Activity and Cognitive Enrichment in Schizophrenia (PACES)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Shaun M. Eack, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19050382; R01MH118267 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Negative Symptoms; Cognition; Social Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This proposed study consists of an 18-month randomized-controlled trial in which 90 outpatients with schizophrenia with moderate-to-severe persistent negative symptoms will be randomized to Cognitive Enhancement Therapy (CET) or Enriched Supportive Therapy (EST) and treated for 18 months. Comprehensive measures of cognition, negative symptoms, and functional outcome will be collected prior to treatment, every 6-months thereafter (6 and 12 months), at treatment completion (18 months), and 3-month (21 months) and one year (30 months) post-treatment follow-up to provide a rigorous confirmatory test of the efficacy of CET and EST for patients with persistent negative symptoms and the cognitive mechanisms of negative symptom improvement in the disorder.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Enhancement Therapy (Experimental): This research treatment aims to help with problems in thinking, planning, and socialization. Participants begin with cognitive training using computer software programs. They also participate in a small social-cognitive group to learn about their condition and how to act wisely in social situations by developing the abilities needed to understand another person's perspective, evaluate social contexts, and be foresightful.
  Time commitment: about 3½ hours per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Enriched Supportive Therapy (Active Comparator): This research treatment uses individual supportive therapy to help patients learn about schizophrenia, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Time commitment: about 2 hours per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Enriched Supportive Therapy

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — An 18-month comprehensive, small group approach for the remediation of cognitive deficits in neurodevelopmental disorders consisting of individual sessions and 45 group training sessions in social cognition that are integrated with approximately 60 hours of computer assisted training in attention, memory, and problem solving skills.
  Other Names: CET
  Arms: Cognitive Enhancement Therapy
Behavioral: Enriched Supportive Therapy — An 18-month intervention that uses individual supportive therapy to help patients learn about schizophrenia, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Other Names: EST
  Arms: Enriched Supportive Therapy

SUMMARY:
This project will conduct a confirmatory efficacy trial of two novel psychosocial interventions, Cognitive Enhancement Therapy and Enriched Supportive Therapy, for the treatment of persistent negative symptoms in schizophrenia.

DETAILED DESCRIPTION:
This project will conduct a confirmatory efficacy trial to examine the efficacy of Cognitive Enhancement Therapy (CET) and Enriched Supportive Therapy (EST) for the treatment of schizophrenia patients with significant and persistent negative symptoms. A total of 90 stabilized schizophrenia outpatients with moderate-to-severe persistent negative symptoms will be randomized to 18 months of CET or EST. Comprehensive data on persistent negative symptoms, social and non-social cognition, and functional outcome will be collected prior to treatment and at frequent 6-month intervals to (1) confirm the efficacy of CET and EST for improving persistent negative symptoms; (2) confirm the impact of cognitive target engagement on reduced negative symptoms; and (3) examine the short-term durability of CET and EST effects on negative symptoms and functioning.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be evaluated longitudinally in a 4-week evaluation period. Patients will be included if they are outpatients and:

1. are between 18-60 years of age;
2. have a diagnosis of schizophrenia or schizoaffective disorder confirmed by the SCID;
3. have a clinical history of persistent negative symptoms lasting at least 3 months as identified from the medical record;
4. have observed persistent negative symptoms at the beginning and end of the 4-week evaluation period;
5. have been stabilized on antipsychotic medication at the beginning and end of the 4-week evaluation period;
6. have stabilized depressive symptoms at the beginning and end of the 4-week evaluation period;
7. have mild or absent extrapyramidal symptoms at the beginning and end of the 4-week evaluation period;
8. have had changes to their primary antipsychotic medication within the previous 3 months;
9. have current IQ > 80; and
10. are able to read (sixth grade level or higher) and speak fluent English. -

Exclusion Criteria:

Exclusion criteria are intended to avoid likely treatment confounders and contraindications and include:

1. the presence of organic brain syndrome;
2. comorbid medical disorders producing cognitive impairment (e.g., mild brain injury, previous concussions with loss of consciousness);
3. persistent suicidal or homicidal behavior;
4. significant clinician-estimated medication non-adherence; and
5. SCID-verified substance use disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Persistent Negative Symptoms | Prior to treatment, 6 months, 12, months, 18 months, 21 months and 30 months
  Negative symptoms will be assessed using the Clinical Assessment Interview for Negative Symptoms (CAINS). The CAINS is a structured interview measure of expressive and motivational negative symptoms consisting of 13 items based on a standardized interview with anchor points for each rating. This measure was developed to address the limitations of previous negative symptom measures and designed for use in clinical trials of negative symptom therapeutics. This outcome has two endpoints that will be evaluated in this trial, persistent negative symptoms related to expression (Expression subscale) and persistent negative symptoms related to motivation/pleasure (Motivation/Pleasure subscale). Items are rated on a 0 to 4 scale, with higher scores indicating greater negative symptom severity.

SECONDARY OUTCOMES:
Change in Functioning | Prior to treatment, 6 months, 12, months, 18 months, 21 months and 30 months
  A composite index of functional outcomes will be derived from measures of social adjustment commonly used in schizophrenia research. These are clinical interview-based measures of functioning, with some self-report measures, covering vocational, social, family, and other functional outcome domains. Measures will include the Social Adjustment Scale-II, Major Role Adjustment Inventory, the Global Assessment of Functioning, and other field standards of functional outcome in schizophrenia. Because these measures do not share a common Unit of Measure and because of the large number of functional outcome measures used, a composite index will be formed to assess changes in functioning to reduce Type I error from multiple inference testing.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed study has a data sharing plan consistent with NIH policy. Data will be de-identified before sharing on a need to know basis. Sharing will be executed with an approved data transfer agreement.
Time Frame: Final data that has not yet been published will be shared after acceptance of publication of the relevant paper.
Access Criteria: Data sharing will occur at two levels:1) specific requests to analyze data from investigators in the field and 2) collaboration with NIH to facilitate data sharing activities for the NIMH National Database for Clinical Trials Related to Mental Illness (NDCT).